CLINICAL TRIAL: NCT07178392
Title: Research on the Disease-syndrome Characteristics of Idiopathic Pulmonary Fibrosis
Brief Title: Disease-syndrome Characteristics of IPF
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Other Study IDs: Characteristics of IPF
Record Dates: First submitted 2025-06-29; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Idiopathic Pulmonary Fibrosis; TCM; Epidemiological investigation; characteristics
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood,Tongue coating
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants fill out the questionnaire: Participants fill out the questionnaire

SUMMARY:
This study, based on previous registration records, aims to explore the syndrome patterns, disease characteristics, and their interrelationships of IPF at different stages, grades, and in its natural course, thus providing a multidimensional interpretation of the syndrome patterns and characteristics of IPF.

DETAILED DESCRIPTION:
This study, based on previous registration records, uses a cross-sectional survey design to collect demographic information, disease-related data, syndrome data, and auxiliary examination data from 2864 IPF patients in China. It aims to elucidate the syndrome types, disease characteristics, and the interrelationships between them of IPF at different stages, grades, and in its natural course.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with IPF;
2. Age ≥ 18 years old;
3. Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients with confusion, dementia, consciousness disorders, and various mental illnesses;
2. Those who are unable to take care of themselves and have been bedridden for a long time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic pulmonary fibrosis (IPF) is a special type of idiopathic interstitial pneumonia, which is mainly manifested by irritating dry cough and progressive dyspnea.
Sampling Method: Non-Probability Sample
Enrollment: 2864 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Disease Stage | Evaluate at baseline.
  Recording the disease staging of IPF patients. According to the Adult Idiopathic Pulmonary Fibrosis (Revised Edition) and Progressive Pulmonary Fibrosis: ATS/ERS/JRS/ALAT Official Clinical Practice Guidelines (2022 Edition), and the Chinese Expert Consensus on the Diagnosis and Treatment of Acute Exacerbation of Idiopathic Pulmonary Fibrosis, the disease staging evaluation of IPF is stable phase or acute exacerbation.
Gender, age and physiologic variables (GAP)stage | Evaluate at baseline.
  Recording the GAP stage of IPF patients. GAP stage is a risk stratification method that quantifies the three core parameters of patients: gender, age, and physiological parameters, by calculating the total score and conducting risk stratification.
Pulmonary function classification | Evaluate at baseline.
  Recording the pulmonary function classification of IPF patients. According to The Expert Consensus on the Diagnostic Criteria for Adult Lung Function in China, pulmonary function classification is divided into mild, moderate, and severe grades.
Natural course | Evaluate at baseline.
  Recording the natural course of IPF patient. According to international research, the natural course of IPF can be divided into stable, slow progression, rapid progression, and recurrent acute exacerbation. The specific criteria are as follows: 1.stable: FVC annual decline<0.13L; 2. stable slow progression: FVC annual decline 0.13L-0.21L; 3. Rapid progress: FVC annual decline>0.21L; 4. Recurrent acute exacerbations: Annual number of acute exacerbations ≥ 1.
The Traditional Chinese Medicine(TCM) Syndromes | Evaluate at baseline.
  Evaluate traditional Chinese medicine syndromes by collecting patients' symptoms, signs, and tongue pulse information.
6 Six Minute Walk Distance(6MWD) | Evaluate at baseline.
  6MWD will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
The 30 - second sit - to - stand test(30s STS) | Evaluate at baseline.
  The 30 second sitting and standing test will be used to evaluate lower limb strength and cardiopulmonary function.
A Tool to Assess Quality of life (ATAQ-IPF) total scores | Evaluate at baseline.
  ATAQ-IPF is currently a specialized scale for evaluating the quality of life, consisting of 13 dimensions and 74 items, with each item scored on a 1-5 scale. The higher the score, the worse the quality of life.
St. George's respiratory questionnaire (SGRQ) total scores | Evaluate at baseline.
  SGRQ is a scale used to evaluate the quality of life of patients, which includes three dimensions: symptoms, mobility, and the impact of disease on daily life, with a total of 50 items. The total score range of SGRQ is usually between 0 and 100, with higher scores leading to poorer quality of life.
Dyspnea | Evaluate at baseline.
  Dyspnea will be assessed by modified Medical Research Council(mMRC) scores. A score of 0-4 will be givenaccording to the degree of immediate dyspnea. A higher score indicates a worse condition.
C-reactive protein (CRP) | Evaluate at baseline.
  The CRP level will be detected by ELISA technology.
Krebs Von den Lungen-6（KL-6） | Evaluate at baseline.
  The KL-6 level will be detected by ELISA technology.
The pulmonary artery systolic pressure(PASP) | Evaluate at baseline.
  The PASP will be measured byechocardiogram.
The diameter of the pulmonary artery | Evaluate at baseline.
  The diameter of the pulmonary artery will be measured byechocardiogram.
Forced vital capacity (FVC) | Evaluate at baseline.
  FVC will be applied to assess pulmonary function.
FVC as the percentage of the predicted value (FVC%) | Evaluate at baseline.
  FVC% will be applied to assess pulmonary function.
Diffusing capacity of the lungs for carbon monoxide (DLCO) | Evaluate at baseline.
  DLCO will be applied to assess pulmonary function.
DLCO as the percentage of the predicted value (DLCO%) | Evaluate at baseline.
  DLCO% will be applied to assess pulmonary function.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China